CLINICAL TRIAL: NCT01809834
Title: Evaluation of Stenfilcon A Versus Etafilcon A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CV-12-57
Record Dates: First submitted 2013-01-17; First posted 2013-03-13 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Etafilcon A (Active Comparator): Each participant was randomized to wear the test lens in one eye and the control lens in the other simultaneously
  Interventions: Device: Stenfilcon A
- Stenfilcon A (Experimental): Each participant was randomized to wear the test lens in one eye and the control lens in the other simultaneously
  Interventions: Device: Etafilcon A

INTERVENTIONS:
Device: Etafilcon A
  Arms: Stenfilcon A
Device: Stenfilcon A
  Arms: Etafilcon A

SUMMARY:
Evaluation of two contact lenses

DETAILED DESCRIPTION:
One week dispensing, investigator-masked, randomized, contralateral study comparing the test lens against the control lens. Each subject will be randomized to wear the test lens in one eye and the control lens in the other eye simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Is correctable to a visual acuity of 20/30 or better (in each eye) with their habitual correction and the assigned study lenses;
* Has astigmatism less than or equal to -1.00D;
* Is an adapted soft contact lens wearer;
* Demonstrates an acceptable fit with the study lenses;
* Has no active anterior segment disease or known ocular disease.

Exclusion Criteria:

* A person will be excluded from the study if he/she:
* Has never worn contact lenses before;
* Has any systemic disease affecting ocular health;
* Is using any systemic or topical medications that will affect ocular health;
* Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses;
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye;
* Has any clinically significant lid or conjunctival abnormalities, neovascularization, corneal scars or corneal opacities;
* Is aphakic;
* Has undergone corneal refractive surgery;
* Is participating in any other type of clinical or research study;
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD., FCO, Principal Investigator — Univeristy of Waterloo, Canada
Locations (1):
- Center for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were determined to be ineligible at the screening visit due to their level of astigmatism
Groups:
- All Participants: Each participant was randomized to wear the test lens in one eye and the control lens in the other simulataneously
  Etafilcon A
  Stenfilcon A
Period: Overall Study
Arm/Group | All Participants
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Each participant was randomized to wear the test lens in one eye and the control lens in the other simultaneously
  Etafilcon A
  Stenfilcon A
Arm/Group | All Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (9.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 43
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 11
Region of Enrollment [Number; unit: participants]
  Canada | 44

OUTCOME MEASURES:

1. Primary Outcome: Participant's Subjective Rating of Comfort (Questionnaire)
Description: Participants rated their comfort of lenses by subjective questionnaire (un-annotated scale, 0-100, 0=Poor comfort/intolerable, 100=Excellent comfort/cannot be felt) Change over time measured at insertion, After settling, 12-hours, 1-week
Time Frame: Insertion, After Lens settling, 12-hours, 1-week
Population: One participant temporarily discontinued from study after 12-hour visit. (n=43 at 1-week visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Etafilcon A; Stenfilcon A: Each participant was randomized to wear the test lens in one eye and the control lens in the other simultaneously
  Etafilcon A
  Stenfilcon A
Arm/Group | Etafilcon A | Stenfilcon A
Number analyzed (Participants) | 44 | 44
Number analyzed (eyes) | 44 | 44
units on a scale
  Insertion | 92 (11) | 91 (11)
  After settling | 96 (7) | 93 (10)
  12-hours | 91 (12) | 88 (13)
  1-week | 90 (10) | 90 (10)

2. Secondary Outcome: Investigator's Objective Assessment of Lens Surface Wettability (Biomicroscopy)
Description: Investigators assigned a lens surface wettability grade by biomicroscopy assessment (grading scale, 0 to 4, 0=excellent, 4=severely reduced).
  Change over time measured after lens settling (insertion), after 12-hours wear on the dispense day (12-hours), after a minimum on one hour of lens wear at 1 week (1-week).
Time Frame: Insertion, 12 hours, 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Etafilcon A | Stenfilcon A
Number analyzed (Participants) | 44 | 44
Number analyzed (eyes) | 44 | 44
units on a scale
  Insertion | 0.69 (0.82) | 0.78 (0.89)
  12-hours | 1.51 (1.26) | 1.47 (1.16)
  1-week | 1.06 (1.00) | 1.15 (0.98)

3. Secondary Outcome: Investigator's Objective Assessment of Overall Fit Acceptance (Biomicroscopy)
Description: Investigators assigned an overall fit acceptance grade by biomicroscopy assessment (grading scale, 0-4, 0=very poor, 4=very good).
  Change over time measured at insertion, 12-hours, 1-week
Time Frame: Insertion, 12 hours, 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Etafilcon A | Stenfilcon A
Number analyzed (Participants) | 44 | 44
Number analyzed (eyes) | 44 | 44
units on a scale
  Insertion | 3.37 (0.47) | 3.44 (0.42)
  12-hours | 3.26 (0.47) | 3.40 (0.37)
  1-week | 3.36 (0.40) | 3.48 (0.31)

4. Primary Outcome: Participant's Subjective Rating of Dryness (Questionnaire)
Description: Participants rated dryness of the lenses by subjective questionnaire (annotated scale, 0-100, 0=cannot be worn / extremely dry, 100=no dryness experienced at any time) Change over time measured at 12-hours, 1-week
Time Frame: 12-hours, 1-week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Etafilcon A | Stenfilcon A
Number analyzed (Participants) | 44 | 44
Number analyzed (eyes) | 44 | 44
units on a scale
  12-hours | 86 (17) | 83 (21)
  1-week | 83 (20) | 82 (21)

5. Primary Outcome: Participant's Subjective Rating of Lens Handling for Insertion (Questionnaire)
Description: Participants rated their lens handling experience for lens insertion by questionnaire (un-annotated scale, 0-100, 0=could not place lens on eye, 100=always easy to place lens on eye) Measured at Dispensing
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Etafilcon A | Stenfilcon A
Number analyzed (Participants) | 44 | 44
Number analyzed (eyes) | 44 | 44
score on a scale | 80 (19) | 86 (14)

6. Primary Outcome: Participant's Subjective Rating of Lens Handling for Removal (Questionnaire)
Description: Participants rated their lens handling experience for the lens removal by questionnaire (un-annotated scale, 0-100, 0=could not remove lens from eye, 100=always easy to remove lens from eye) Change over time measured at 12-hours, 1-week
Time Frame: 12-hours, 1-week
Population: One participant temporarily discontinued from study after 12-hour visit. (n=43 at 1-week visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Etafilcon A | Stenfilcon A
Number analyzed (Participants) | 44 | 44
Number analyzed (eyes) | 44 | 44
units on a scale
  12-hours | 97 (7) | 92 (15)
  1-week | 94 (12) | 94 (9)

7. Primary Outcome: Participant's Subjective Rating of Visual Quality (Questionnaire)
Description: Participants rated visual quality of the lenses by questionnaire (annotated scale, 0-100, 0=extremely poor vision all of the time. Cannot function, 100=excellent vision all of the time) Change over time measured at 12-hours, 1-week
Time Frame: 12-hours, 1-week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Etafilcon A | Stenfilcon A
Number analyzed (Participants) | 44 | 44
Number analyzed (eyes) | 44 | 44
units on a scale
  12-hours | 92 (13) | 89 (15)
  1-week | 89 (12) | 89 (14)

8. Primary Outcome: Participant's Subjective Rating of Overall Preference (Questionnaire)
Description: Participants rated their overall lens preference by questionnaire. (annotated scale, 0-100, scale normalized to 0=no preference, +50=strongly prefers test lens, -50=strongly prefers control lens). Change over time measured at 12-hours, 1-week
Time Frame: 12-hours, 1-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 44
score on a scale
  12-hours | -8 (24)
  1-week | 5 (16)

9. Secondary Outcome: Investigator's Objective Assessment of Visual Acuity, High Contrast at High Illumination (Snellen)
Description: Investigators tested participants using snellen charts distant to the participant in each eye (monocular) at normal lighting conditions (high illumination).
  (logMAR, 0.00 = 20/20 Snellen acuity, positive values = poorer visual acuity, negative values = better visual acuity). Change over time measured at insertion, 12-hours, 1-week.
Time Frame: Insertion
Measure: Log Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Etafilcon A | Stenfilcon A
Number analyzed (Participants) | 44 | 44
Number analyzed (eyes) | 44 | 44
logMAR
  Insertion | -0.09 (0.09) | -0.08 (0.08)
  12-hours | -0.09 (0.07) | -0.08 (0.07)
  1-week | -0.09 (0.06) | -0.08 (0.07)

10. Secondary Outcome: Investigator's Objective Assessment of Visual Acuity, High Contrast at Low Illumination (Snellen)
Description: Investigators tested participants using snellen charts distant to the participant in each eye (monocular) at low lighting conditions (low illumination).
  (logMAR, 0.00 = 20/20 Snellen acuity, positive values = poorer visual acuity, negative values = better visual acuity). Change over time measured at insertion, 12-hours, 1-week.
Time Frame: Insertion, 12-hours, 1-week
Measure: Log Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Etafilcon A | Stenfilcon A
Number analyzed (Participants) | 44 | 44
Number analyzed (eyes) | 44 | 44
logMAR
  Insertion | -0.07 (0.08) | -0.06 (0.07)
  12-hours | -0.07 (0.07) | -0.07 (0.07)
  1-week | -0.08 (0.07) | -0.07 (0.07)

11. Secondary Outcome: Investigator's Objective Assessment of Anterior Ocular Physiological Response, Cornea (Biomicroscopy)
Description: Investigators assigned an anterior ocular physiological response grade by biomicroscopy assessment with corneal staining (grading scale, 0-4, 0=none, 4=severe) Change over time measured at baseline (screening and dispensing visit), 12-hours, 1-week
Time Frame: Baseline, 12-hours, 1-week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Etafilcon A | Stenfilcon A
Number analyzed (Participants) | 44 | 44
Number analyzed (eyes) | 44 | 44
units on a scale
  baseline Central | 0.08 (0.28) | 0.23 (0.48)
  baseline Nasal | 0.47 (0.67) | 0.56 (0.74)
  baseline Temporal | 0.23 (0.61) | 0.14 (0.38)
  baseline Superior | 0.30 (0.60) | 0.25 (0.51)
  baseline Inferior | 0.70 (0.97) | 0.55 (0.70)
  12-hours Central | 0.08 (0.26) | 0.16 (0.44)
  12-hours Nasal | 0.09 (0.31) | 0.32 (0.66)
  12-hours Temporal | 0.24 (0.61) | 0.16 (0.40)
  12-hours Superior | 0.23 (0.45) | 0.32 (0.51)
  12-hours Inferior | 0.68 (0.89) | 0.74 (0.87)
  1-week Central | 0.10 (0.35) | 0.12 (0.39)
  1-week Nasal | 0.23 (0.51) | 0.24 (0.48)
  1-week Temporal | 0.22 (0.51) | 0.16 (0.41)
  1-week Superior | 0.17 (0.44) | 0.23 (0.54)
  1-week Inferior | 0.69 (0.74) | 0.51 (0.82)

12. Secondary Outcome: Investigator's Objective Assessment of Anterior Ocular Physiological Response, Conjunctiva (Biomicroscopy)
Description: Investigators assigned an anterior ocular physiological response grade by biomicroscopy assessment with conjuncitval staining (grading scale, 0-4, 0=none, 4=severe) Change over time measured at baseline (screening and dispensing visit), 12-hours, 1-week
Time Frame: Baseline, 12-hours, 1-week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Etafilcon A | Stenfilcon A
Number analyzed (Participants) | 44 | 44
Number analyzed (eyes) | 44 | 44
units on a scale
  baseline Nasal | 0.23 (.035) | 0.21 (0.38)
  baseline Temporal | 0.15 (0.25) | 0.11 (0.21)
  baseline Superior | 0.06 (0.19) | 0.06 (0.19)
  baseline Inferior | 0.09 (0.29) | 0.08 (0.26)
  12-hours Nasal | 0.86 (0.73) | 0.72 (0.57)
  12-hours Temporal | 0.55 (0.55) | 0.93 (0.59)
  12-hours Superior | 0.17 (0.24) | 0.59 (0.73)
  12-hours Inferior | 0.63 (0.74) | 0.76 (0.68)
  1-week Nasal | 0.83 (0.62) | 0.52 (0.56)
  1-week Temporal | 0.34 (0.41) | 0.55 (0.57)
  1-week Superior | 0.17 (0.30) | 0.33 (0.44)
  1-week Inferior | 0.65 (0.85) | 0.50 (0.66)

ADVERSE EVENTS:
Groups:
- All Participants: Each participant was randomized to wear the test lens in one eye and the control lens in the other
  Etafilcon A
  Stenfilcon A
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

LIMITATIONS AND CAVEATS:
One participant temporarily discontinued after 12-hour visit. (Primary outcome 1 and 4,1-week visit, n=43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less